CLINICAL TRIAL: NCT00302224
Title: A Phase 1/2a, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Study of Safety, Tolerability, Pharmacokinetics and Activity of 14 Days of Oral Dosing With the 2S,4R Enantiomer of Ketoconazole (DIO-902) in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Phase 1/2a Study of the 2S,4R Enantiomer of Ketoconazole in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DiObex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIO-501
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Type 2 Diabetes
Keywords: safety; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: 2S, 4R Ketoconazole (DIO-902)

SUMMARY:
The study is designed to test the safety, tolerability of a newly developed form of ketoconazole (DIO-902) for the treatment of elevated blood sugars in type 2 diabetes. This study also will also examine the effect of the drug on total and LDL cholesterol and blood pressure. Elevated cortisol may contribute to the development of Type II diabetes. The investigational drug DIO-902 may reduce the level of cortisol in blood and therefore provide better control of blood sugar levels in patients with Type II diabetes.

DETAILED DESCRIPTION:
DiObex is developing a modified form of ketoconazole (enantiomer) (DIO-902) as an investigational new drug for the treatment of the elevated blood sugar associated with type 2 diabetes. Other benefits may include reduced total and LDL cholesterol, and reduced blood pressure. With chronic treatment, reduced visceral fat may also be seen. Ketoconazole (racemic) is an approved drug for the treatment of a variety of fungal infections. The approved racemic ketoconazole inhibits cortisol synthesis. In patients with Cushings Disease racemic ketoconazole reduces glucose, cholesterol and blood pressure. Elevated cortisol may be a contributing causal factor in the development of type 2 diabetes; clinical trials with racemic ketoconazole have been carried out in these patients. The results of these clinical trials support the concept of treating type 2 diabetes through a lowering of plasma cortisol and provide evidence of the safety and tolerability of racemic ketoconazole. Racemic ketoconazole has, however, been associated with liver toxicity which is generally mild in nature. However, in rare cases (1:10,000 to 15,000 patients) severe liver toxicity may occur, and in extremely rare cases this adverse event may be irreversible and life-threatening. Preclinical results suggest that DIO-902 may be both safer and more efficacious than the racemic mixture.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 70
2. Females are non-lactating and using adequate contraception, in the opinion of the Principal Investigator and negative serum pregnancy test if of child bearing potential (intact uterus and pre-menopausal)
3. Diagnosis of type 2 diabetes mellitus (DM) for at least 6 months. Type 2 diabetes may be untreated or may be treated with diet and exercise only and/or pharmacologic therapy as in Inclusion Criterion 4
4. Pharmacologic treatment for type 2 DM may include the following and must be stable for > 3 months Glucophage (Metformin) (< maximum dose of 2550 mg) or Glucophage XR (< maximum dose of 2000 mg)
5. HbA1C level of 6.5 to 10.9%
6. Fasting C-peptide level of greater than or equal to 0.8 nmol/L (2.4 ng/mL)
7. ACTH stimulation test results with any cortisol level (baseline, 30 or 60 minutes) of >18 µg/dL
8. Normal thyroid stimulating hormone

9.12-lead electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality

10.BMI of 26 to 40 kg/m2

11.Subjects with a history of hypertension may be on a stable anti-hypertensive regimen (except those drugs stated under Exclusion Criterion 7) for > 2 months

12.Ability to comprehend and a willingness to provide informed consent

Exclusion Criteria:

1. History of any atherosclerotic disorder (myocardial infarction, angina, cerebrovascular accident, peripheral vascular disease or congestive heart failure secondary to ischemic myocardial injury) that would, in the estimation of the Investigator, make it unsafe to stop all lipid lowering drugs during the course of the study
2. Known hypersensitivity or idiosyncratic reaction related to ketoconazole or other imidazole compounds
3. History of malignancy (except basal cell carcinoma) within the 3 years before the initial dose of the study medication
4. Excessive alcohol intake or drug abuse using the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV), criteria
5. Any other clinically significant medical condition, as determined by the Investigator. These clinically significant medical conditions include proliferative diabetic retinopathy and neuropathic symptoms that limit activities of daily living
6. Participation in another clinical trial and/or treatment received with any investigational agent within one month before the initial dose of study medication
7. Concomitant therapy with the following: any antacid or ulcer medication, weight loss medications, oral or injected hypoglycemics (metformin is allowed) or insulin, steroids, cyclosporine, tacrolimus, midazolam, digoxin, coumarin derivatives, phenytoin, rifampin, loratadine, HIV protease inhibitors, spironolactone, thiazide diuretics, calcium channel blockers and erythromycin. Subjects taking lipid lowering medications may be enrolled if Investigator determines that subject does not have any conditions that preclude this cessation and subject is willing to stop such medications 21 days prior to Study Visit 1 through Study Visit 3 (Day 16)
8. History of HIV
9. Positive hepatitis B (HBsAg) or positive hepatitis C (Hepatitis C antibody) test during Screening
10. WBC count <4000/µL or >14,000/µL
11. Hemoglobin <12.0 gm/dL in females and <14.0 gm/dL in males
12. Any single hepatic enzyme (ALT, AST, AP and total bilirubin) is greater than the upper limit of the normal reference range used by the central laboratory
13. Creatinine > 1.5 times the upper limit of normal
14. Known hypersensitivity to cosyntropin (ACTH) or any component of the formulation (mannitol or sodium chloride)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02; Study Completion 2006-08

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of 14 daily doses; To determine the pharmacokinetic (PK) profile in plasma of DIO-902 after a single dose, and after fourteen daily doses; To evaluate the pharmacodynamic effects of fourteen daily doses

SECONDARY OUTCOMES:
To explore the impact of treatment with the enantiomer of ketoconazole on markers of inflammation and coagulation as well as on lipomic profiles, pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Schwartz, MD, Principal Investigator — Diabetes and Glandular Disease Clinic
Locations (5):
- United States (5):
  - Asha Thomas, MD - Medstar, Washington D.C., District of Columbia
  - Marc Rendell, MD - Creighton University, Omaha, Nebraska
  - Dr. Andrew Ahmann, MD - Radiant Research, Portland, Oregon
  - Carlos Arauz-Pacheco, MD - Radiant Research, Dallas, Texas
  - Sherwin Schwartz, MD - Diabetes and Glandular Disease Clinic, San Antonio, Texas